CLINICAL TRIAL: NCT07094737
Title: The ITACARE-P CardioRehab Registry
Brief Title: The Italian Alliance for Cardiovascular Rehabilitation and Prevention (ITACARE-P) Registry: An Observational Study on Cardiac Rehabilitation in Patients With Coronary Disease or Heart Failure
Acronym: CardioRehab
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); ASST Crema (Unknown); IRCCS Ospedale San Raffaele (Other); AORN Sant'Anna e San Sebastiano - Caserta (Unknown); IRCCS Fondazione Don Gnocchi-Firenze (Unknown); Fondazione Don Gnocchi Parma (Unknown); U.O.S. Riabilitazione Cardiologica Area Sud Azienda USL Toscana (Unknown); S.O.D. Riabilitazione Cardiologica Azienda Ospedaliero Universitaria Careggi Firenze (Unknown); UOSD Cardiologia Riabilitativa Azienda Ospedaliera San Giovanni-Addolorata (Unknown); IRCCS Istituti clinici Maugeri, Istituto di Montescano (Unknown); IRCCS Istituti clinici Maugeri, Istituto di Pavia (Unknown); IRCCS Istituti clinici Maugeri, Istituto di Gattico-Veruno (Unknown); Struttura complessa Riabilitazione Cardiologica (Unknown); Casa di cura villa gemma (Unknown); Cardiologia Riabilitativa Tagliacozzo (Unknown); ASST Brianza (Unknown); Riabilitazione del Cardiopatico (Unknown); UOS Cardiologia Riabilitativa ULSS Serenissima (Unknown); Ospedale Riabilitativo di Alta Specializzazione (Unknown); Istituto clinico Maugeri Lumezzane (Unknown); U.O.C. Cardiologia ASL 3 Genovese (Unknown)
Responsible Party: Sponsor
Other Study IDs: CardioRehab
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Rehab; Heart Failure; Coronary Disease; Heart Conditions; Rehabilitation; Cardiac Rehabilitation; Telerehabilitation
Keywords: Cardiac Rehab; Heart Failure; Coronary disease; Heart conditions; Rehabilitation; Cardiac rehabilitation; Telerehabilitation
MeSH Terms: conditions — Heart Failure; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiorehab patients: cardiological rehabilitation patients with heart conditions (heart coronary deseases and/or heart failure).

SUMMARY:
ITACARE-P CardioRehab Registry is a nationwide observational study conducted in Italy and coordinated by the Fondazione Don Carlo Gnocchi in Milan. It involves multiple hospitals and rehabilitation centers across the country and aims to better understand how cardiac rehabilitation (CR) is delivered to patients recovering from heart conditions (coronary deseases and/or heart failure). CR is a structured program that includes exercise, lifestyle education, and psychological support, and is known to improve recovery, reduce future cardiac events, lower hospital readmissions, and enhance quality of life. Despite strong recommendations from international guidelines, not all eligible patients are referred to CR, and its delivery varies. This study collects real-world data to describe how CR programs are implemented, evaluate patient outcomes, identify subgroups needing tailored care, and support improvements in cardiac care services in Italy. Adults who recently experienced a qualifying heart condition are enrolled and followed during their standard rehabilitation, without any changes to treatment. Data on medical history, risk factors, quality of life, functional improvements, and medication use are collected, with follow-up at 6 and 12 months. Participation involves no added risks, and personal health data is securely managed according to EU GDPR regulations using the REDCap system. The study aims to enhance the quality, consistency, and equity of cardiac rehabilitation across the country.

DETAILED DESCRIPTION:
The ITACARE-P CardioRehab Registry, is a nationwide observational project conducted in Italy. It is led by the Fondazione Don Carlo Gnocchi in Milan and involves several hospitals and rehabilitation centers across all the Country.

The main goal of the present study is to better understand how cardiac rehabilitation (CR) is being delivered to patients who have experienced heart-related conditions (coronary deseases or heart failure). Cardiac rehabilitation is a structured program that includes exercise, lifestyle education, and psychological support. It is known to help patients recover faster, reduce the risk of future heart problems, lower hospital readmissions, and improve quality of life.

Despite strong recommendations from international guidelines, not all eligible patients are referred to cardiac rehabilitation, and CR programs are not always delivered in a consistent way. This study aims to collect real-world data to:

* Describe how CR programs are implemented in different hospitals,
* Evaluate whether patients are meeting treatment goals (such as improved fitness, lower cholesterol, or better medication use),
* Identify patient groups that may need different types of care,
* Support future improvements in heart care services in Italy and beyond.

The central idea behind the study is that systematically collecting and analyzing data on patients undergoing cardiac rehabilitation can highlight what works best, help standardize care, and improve long-term health outcomes for people with heart disease. By understanding how care is delivered and what results are achieved, the study aims to improve the quality and equity of cardiac rehabilitation services across Italy.

Adults who recently had a heart condition that qualifies them for cardiac rehabilitation will be included.

This is not a treatment trial, and no experimental therapies are given. Instead, the study observes what happens during standard care. Patients will continue to receive their normal rehabilitation program/care. Information will be collected about:

Basic personal and medical data (such as age, blood pressure, cholesterol),

Risk factors (like smoking, diabetes, weight),

Emotional well-being and quality of life,

Functional improvements (like exercise capacity),

Medication use.

Patients will also be contacted by phone at 6 and 12 months after their program to check on their health and whether they have had any additional heart-related problems.

There are no added risks because this study does not involve any changes to a patient's usual care. While there are no direct personal benefits, participants may experience better tracking of their health indicators. More importantly, their participation helps researchers and healthcare providers improve care for future patients.

All personal health data will be kept confidential and protected according to European Union data protection regulations (GDPR). A secure online system (REDCap) will be used to collect and manage the data. The information will be pseudo-anonymized, meaning names and personal identifiers will ben removed, so no one can be identified and only authorized staff will have access to the data and it will only be used for scientific and quality improvement .

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease and/or heart failure who meet the current regulatory requirements for appropriateness of referral to cardiac rehabilitation are eligible for enrollment. These patients may be included regardless of whether they are referred to inpatient or outpatient cardiac rehabilitation programs, depending on the clinical setting and care pathway.

Exclusion Criteria:

* Explicit refusal to participate in the study by the patient;
* Planned hospital readmission within six months after completion of the cardiac rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiological rehabilitation patients with heart conditions (heart coronary deseases and/or heart failure).
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of mace in cardiorehab population | 6 months and 12 months
  Evaluate how cardiac rehabilitation (CR) is delivered across Italy and to assess its real-world effectiveness in patients recovering from major cardiovascular events such as coronary deseases or heart failure. A key focus of the study is to measure the incidence of major adverse cardiovascular events (MACE)-including cardiovascular death, recurrent myocardial infarction, stroke, and hospital readmissions-during a 12-month follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Dongnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No